CLINICAL TRIAL: NCT06788756
Title: A Pivotal Phase 2/3, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Adaptive Design Study of L Annamycin for Injection in Combination With Cytarabine Injection Versus Placebo in Combination With Cytarabine Injection as Second Line Therapy for Remission Induction in Adult Subjects With Refractory/Relapsed Acute Myeloid Leukemia
Brief Title: L-Annamycin for Injection in Combination With Cytarabine Injection as Second Line Therapy for Remission Induction in Adult Subjects With Refractory/Relapsed AML
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Moleculin Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: MB-108; 2024-518359-47-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-05; First posted 2025-01-23 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukaemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Part A / Treatment Arm 1 (Placebo Comparator): placebo (0.9% Sodium Chloride Injection, i.e., the diluent for L-Annamycin for Injection) for three consecutive days in combination with 2.0 g/m2/day Cytarabine Injection for five consecutive days
  Interventions: Drug: Placebo in combination with Cytarabine Injection
- Part A / Treatment Arm 2 (Active Comparator): 190 mg/m2/day L-Annamycin for Injection for three consecutive days in combination with 2.0 g/m2/day Cytarabine Injection for five consecutive days.
  Interventions: Drug: Liposomal Annamycin Injection in combination with Cytarabine Injection
- Part A / Treatment Arm 3 (Active Comparator): 230 mg/m2/day L-Annamycin for Injection for three consecutive days in combination with 2.0 g/m2/day Cytarabine Injection for five consecutive days.
  Interventions: Drug: Liposomal Annamycin Injection in combination with Cytarabine Injection
- Part B / Treatment Arm 1 (Placebo Comparator): Placebo (0.9% Sodium Chloride Injection) for three consecutive days in combination with 2.0 g/m2/day Cytarabine Injection for five consecutive days (i.e., the same as Treatment Arm 1 of Part A).
  Interventions: Drug: Placebo in combination with Cytarabine Injection
- Part B / Treatment Arm X (Active Comparator): Optimal dosage regimen (as determined in Part A) of L Annamycin for Injection (190 mg/m2/day or 230 mg/m2/day) for three consecutive days in combination with 2.0 g/m2/day Cytarabine Injection for five consecutive days (i.e., the same as Treatment Arm 2 or 3, respectively, of Part A).
  Interventions: Drug: Liposomal Annamycin for Injection in combination with Cytarabine Injection.

INTERVENTIONS:
Drug: Placebo in combination with Cytarabine Injection — placebo (0.9% Sodium Chloride Injection, i.e., the diluent for L-Annamycin for Injection) for three consecutive days in combination with 2.0 g/m2/day Cytarabine Injection for five consecutive days.
  Arms: Part A / Treatment Arm 1; Part B / Treatment Arm 1
Drug: Liposomal Annamycin Injection in combination with Cytarabine Injection — 190 mg/m2/day L-Annamycin for Injection for three consecutive days in combination with 2.0 g/m2/day Cytarabine Injection for five consecutive days.
  Arms: Part A / Treatment Arm 2
Drug: Liposomal Annamycin Injection in combination with Cytarabine Injection — 230 mg/m2/day L-Annamycin for Injection for three consecutive days in combination with 2.0 g/m2/day Cytarabine Injection for five consecutive days.
  Arms: Part A / Treatment Arm 3
Drug: Liposomal Annamycin for Injection in combination with Cytarabine Injection. — optimal dosage regimen (as determined in Part A) of L Annamycin for Injection (190 mg/m2/day or 230 mg/m2/day) for three consecutive days in combination with 2.0 g/m2/day Cytarabine Injection for five consecutive days (i.e., the same as Treatment Arm 2 or 3, respectively, of Part A).
  Arms: Part B / Treatment Arm X

SUMMARY:
This pivotal phase 2/3, multi-center, adaptive design study of L-Annamycin for Injection in combination with Cytarabine Injection as second line therapy for remission induction in adult subjects with refractory/relapsed AML is divided into two parts, Part A and Part B.

DETAILED DESCRIPTION:
This pivotal phase 2/3, multi-center, adaptive design study of L-Annamycin for Injection in combination with Cytarabine Injection as second line therapy for remission induction in adult subjects with refractory/relapsed AML is divided into two parts, Part A and Part B.

Part A (Determination of Optimal Dosage Regimen) Part A of this study is a randomized, double-blind, placebo-controlled (RDBPC), efficacy, safety, tolerability, and pharmacokinetics study comparing two dose levels of L Annamycin for Injection (190 versus 230 mg/m2/day) in combination with Cytarabine Injection (2.0 g/m2/day) versus placebo in combination with Cytarabine Injection to identify the optimal dosage regimen as second line therapy for remission induction in adult subjects with refractory/relapsed AML.

Seventy-five to ninety subjects with a pathologically confirmed diagnosis of AML who have refractory/relapsed AML after having received only one prior line of therapy will be enrolled in Part A. A prior line of therapy will be defined as the planned therapy consisting of one or more cycles of episodic treatment or a defined period of continuous treatment. This may consist of single-agent or combination therapy as well as a planned sequence of treatment phases. For example, first-line treatment of AML with induction, consolidation, and allogeneic hematopoietic stem cell transplantation (alloHSCT) is considered one line of therapy. A line of therapy ends when the patient fails to achieve a response within a prespecified period (refractory) or relapses after achieving CR. For the purpose of confirming refractory AML at screening, refractory disease will be defined as CR not being achieved after first line therapy [i.e., after 1 cycle of intensive therapy or 180 days after commencing less-intensive therapy (shorter durations of less-intensive therapy may be considered for refractory disease on a case by case basis after discussion between the PI and Medical Monitor)]. Subjects who meet all eligibility criteria after the completion of both screening and baseline assessments will be enrolled. Initially, 45 subjects will be randomized 1:1:1 to one of the three treatment arms listed below (i.e.,approximately 15 per treatment arm). Randomization will be stratified by continent. Depending on the outcome of the first interim analysis (see further below), additional subjects will either be randomized 1:1:1 to one of the three treatment arms listed below (for a total of approximately 30 per treatment arm in Part A) randomized 1:1 to either placebo in combination with Cytarabine Injection (Treatment Arm 1) or the L-Annamycin for Injection in combination with Cytarabine Injection arm that was selected to continue after the first interim analysis (i.e., Treatment Arm 2 or 3) (for a total of approximately30 per treatment arm in Part A, except for the arm that is dropped after the first interim analysis, which will have a total of approximately ≤15 and ≤30, depending on how many subjects were enrolled at the point the decision to drop the arm occurs).

* Treatment Arm 1: placebo (0.9% Sodium Chloride Injection, i.e., the diluent for L-Annamycin for Injection) for three consecutive days in combination with 2.0 g/m2/day Cytarabine Injection for five consecutive days.
* Treatment Arm 2: 190 mg/m2/day L-Annamycin for Injection for three consecutive days in combination with 2.0 g/m2/day Cytarabine Injection for five consecutive days.
* Treatment Arm 3: 230 mg/m2/day L-Annamycin for Injection for three consecutive days in combination with 2.0 g/m2/day Cytarabine Injection for five consecutive days.

L-Annamycin for Injection will be administered as an intravenous (IV) infusion over 2 hours. The placebo will be administered the same (i.e., IV infusion over 2 hours). Cytarabine Injection will be administered as an IV infusion over 4 hours. The first day of Cytarabine Injection treatment will start on the first day of L-Annamycin for Injection or placebo treatment (Day 1). On the days where both Cytarabine Injection and L-Annamycin for Injection or placebo are administered, the Cytarabine Injection infusion will be initiated after the L-Annamycin for Injection or placebo infusion is completed.The recommended time between infusions is 15 minutes (± 5 minutes). Part A of this study will include two interim analyses as follows:

First Interim Analysis: After the 45 subjects enrolled in Part A of this study have completed their first treatment cycle response assessment at Day 35 ± 14 days, the data for those subjects will be verified/cleaned and locked, and the data will be unblinded and analyzed (n = approximately 15 per treatment arm). Enrollment in the study will not be halted while the first interim analysis is performed. Comparisons will be made between the three treatment arms to determine if continuation of the study should be halted due to a lack of efficacy difference between the placebo in combination with Cytarabine Injection arm (Treatment Arm 1) and the L-Annamycin for Injection in combination with Cytarabine Injection arms (Treatment Arms 2 and 3; i.e., futility analysis) or too excessive of a risk of serious adverse events (SAEs) with Treatment Arms 2 and/or 3 relative to Treatment Arm 1. An unblinded independent data monitoring committee (iDMC) will review the available efficacy, safety, and pharmacokinetic (PK) data and make recommendations to the Sponsor on how to proceed with the remainder of Part A of the study. The primary options will be to recommend that the study be halted for futility reasons, for safety reasons, or that the study continue. If the iDMC recommends that the study continues, they will recommend if one or both L-Annamycin for Injection dosage regimens (i.e., 190 mg/m2/day or 230 mg/m2/day) continue for Part A.

In the European Union (EU), the iDMC recommendations from the first interim analysis will be provided to the Competent Authorities of EU Member States concerned, and if a protocol amendment is needed, it will be submitted within a Substantial Modification.

Second Interim Analysis: After all subjects enrolled in Part A of this study (total of 75 to 90 subjects; see above for explanation of variable total subject number) have completed their first treatment cycle response assessment at Day 35 ± 14 days, enrollment in the study will be temporarily halted, the data will be verified/cleaned and locked, the data for the second group of subjects (i.e., who were not part of the first interim analysis) will be unblinded, and the pooled Part A data will be analyzed. If all three arms were continued after the first interim analysis, three treatment arms will be compared (n = approximately 30 per treatment arm) to determine which of the L Annamycin for Injection dosage regimens (190 mg/m2/day versus 230 mg/m2/day) is the optimal dosage regimen for continuing with for the remainder of the study (Part B) and which dosage regimen will be dropped from further enrollment. If one of the two L Annamycin for Injection in combination with Cytarabine Injection dosage regimens (Treatment Arm 2 or 3) was dropped after the first interim analysis, the remaining arm will be compared against placebo in combination with Cytarabine Injection (Treatment Arm 1) (n = approximately 30 per treatment arm) to confirm that the study should continue with that regimen to Part B.

Part B (Expansion at Optimal Dosage Regimen) Part B of this study is a RDBPC, efficacy, safety, tolerability, and pharmacokinetics study of the optimal dosage regimen of L-Annamycin for Injection in combination with Cytarabine Injection (as determined in Part A) versus placebo in combination with Cytarabine Injection as second line therapy for remission induction in adult subjects with refractory/relapsed AML.

Once the optimal dosage regimen is determined (see Part A above), enrollment will resume under Part B of the study. Approximately 222 additional subjects with a pathologically confirmed diagnosis of AML who have refractory/relapsed AML after having received only one prior line of therapy (i.e., the same patient population as for Part A) will be enrolled in Part B.

Subjects who meet all eligibility criteria after the completion of both screening and baseline assessments will be enrolled and randomized 1:1 to one of the two treatment arms listed below (i.e., 111 per treatment arm). Randomization will be stratified by continent.

* Treatment Arm 1: placebo (0.9% Sodium Chloride Injection) for three consecutive days in combination with 2.0 g/m2/day Cytarabine Injection for five consecutive days (i.e., the same as Treatment Arm 1 of Part A).
* Treatment Arm X: optimal dosage regimen (as determined in Part A) of L Annamycin for Injection (190 mg/m2/day or 230 mg/m2/day) for three consecutive days in combination with 2.0 g/m2/day Cytarabine Injection for five consecutive days (i.e., the same as Treatment Arm 2 or 3, respectively, of Part A).

ELIGIBILITY:
Inclusion Criteria:

1. Has a pathologically confirmed diagnosis of AML per the 2022 International Consensus Classification (ICC) as adopted in the European LeukemiaNet (ELN) 2022 recommendations for the diagnosis and management of AML. The tests and procedures used to establish the diagnosis of AML should be consistent with the ELN's 2022 recommendations
2. Has refractory/relapsed AML after having received only one prior line of therapy*.

   *A prior line of therapy will be defined as the planned therapy consisting of one or more cycles of episodic treatment or a defined period of continuous treatment. This may consist of single-agent or combination therapy as well as a planned sequence of treatment phases. For example, first-line treatment of AML with induction, consolidation, and alloHSCT is considered one line of therapy. A line of therapy ends when the patient fails to achieve a response within a prespecified period (refractory) or relapses after achieving CR. For the purpose of confirming refractory AML at screening, refractory disease will be defined as CR not being achieved after first line therapy [i.e., after 1 cycle of intensive therapy or 180 days after commencing less-intensive therapy (shorter durations of less-intensive therapy may be considered for refractory disease on a case by case basis after discussion between the PI and Medical Monitor)].
3. Between 18 and 80 years of age (inclusive) at the time of signing the informed consent form (ICF).
4. Has received no chemotherapy, radiation, or major surgery within 2 weeks prior to the first randomized dose of study drug or has recovered from the toxic side effects of that therapy. Hydroxyurea to control white blood cell (WBC) count, supportive measures, and prophylaxes as required under the protocol will be allowed. Treatment of opportunistic or other infections with antibiotics, antifungals, and/or antiviral agents, including therapy for meningeal disease (i.e., intrathecal chemotherapy), per institutional standards of care will be allowed during this period, as long as the symptoms of infection have resolved by 1 week prior to the first dose of randomized study drug.
5. Has received no investigational therapy within 4 weeks prior to the first randomized dose of study drug.
6. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 at screening.
7. Has a life expectancy of greater than six weeks at screening.
8. Has adequate laboratory results at screening including the following:

   1. Total bilirubin ≤2.0 times the upper limit of normal (ULN). For subjects with leukemic involvement or Gilbert Syndrome, total bilirubin must be ≤3.0 ULN.
   2. Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase <3.5 times the ULN. For subjects with organ involvement, AST, ALT, and alkaline phosphatase must be ≤4.5 times the ULN.
   3. Creatinine clearance ≥60 mL/min (using Cockcroft-Gault equation).
9. Can understand and sign the ICF, can communicate with the PI, and can understand and comply with the requirements of the protocol.
10. For women of childbearing potential (WCBP): Must have a negative serum beta human chorionic gonadotropin (ß-hCG) pregnancy test within 72 hours prior to the first randomized dose of study drug.
11. For WCBP: Must agree to not donate ova and use a highly effective method of birth control from the time of informed consent through 6 months after their last randomized dose of study drug.
12. For males with partners who are WCBP: Must agree to not donate sperm and use a highly effective method of birth control from the time of informed consent through 6 months after their last randomized dose of study drug.

Exclusion Criteria:

1. Has prior or current diagnosis of acute promyelocytic leukemia (APL) or myelodysplastic syndrome (MDS)/AML
2. Received prior mediastinal radiotherapy.
3. Has central nervous system involvement.
4. Has impaired cardiac function, including any of the following:

   1. Abnormal LVEF at screening [per American College of Cardiology, normal LVEF is 50 to 70%
   2. Valvular heart disease.
   3. Severe, uncontrolled hypertension.
   4. Uncontrolled cardiac arrhythmias.
   5. Recent (≤6 months prior to screening) myocardial infarction.
   6. Unstable angina.
   7. Symptomatic congestive heart failure.
   8. New York Heart Association (NYHA) classification of 3 or 4.
   9. QT interval/corrected QT (QTc) interval >480 msec at screening.
   10. History of additional risk factors for torsade des pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
   11. Use of concomitant medications that significantly prolong the QT/QTc interval.
5. Has clinically relevant serious comorbid medical conditions including, but not limited to, active infection, chronic obstructive or chronic restrictive pulmonary disease, history of positive status for human immunodeficiency virus (virus detected in serum) hepatitis B or hepatitis C with current serious symptoms or signs of underlying chronic infection or psychiatric illness/social situations that would limit compliance with study requirements.
6. Has evidence of mucositis/stomatitis at screening or baseline, or has history of severe (≥Grade 3) mucositis/stomatitis from prior therapy.
7. Has any condition that, in the opinion of the PI, places the subject at unacceptable risk if he/she were to participate in the study.
8. Has received prior treatment with L-asparaginase.
9. Pregnant or breastfeeding.
10. Known hypersensitivity to anthracyclines, cytarabine, the excipients of L Annamycin for Injection or Cytarabine Injection, or contrast media that may be used for the protocol-specified GLS assessments.
11. Has received a total cumulative prior anthracycline dose of > 300 mg/m2 (daunorubicin equivalent dose).
12. Has relapsed or refractory AML with a FLT3 mutation, unless resides in a country where gilteritinib is not available.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Part A -Determination of Optimal Dosage Regimen | From initiation of the first randomized treatment cycle until the first post treatment bone marrow assessment, assessed up to Day 49
  1. To identify the optimal dosage regimen of L Annamycin for Injection (190 versus 230 mg/m2/day) in combination with Cytarabine Injection (2.0 g/m2/day) as second line therapy for remission induction in adult subjects with refractory/relapsed acute myeloid leukemia (AML) as measured by rate of complete remission (CR) after one treatment cycle.
Part B - Expansion at Optimal Dosage Regimen | From initiation of the first randomized treatment cycle until the first post treatment bone marrow assessment, assessed up to Day 49
  To confirm the superior efficacy of the optimal dosage regimen of L-Annamycin for Injection in combination with Cytarabine Injection (determined in Part A) versus placebo in combination with Cytarabine Injection as second line therapy for remission induction in adult subjects with refractory/relapsed AML as measured by rate of CR after one treatment cycle

SECONDARY OUTCOMES:
Part A -Comparison of Efficacy as Measured by Overall Survival (OS) | From date of randomization to treatment (Day 1) to the date of death from any cause, assessed up to 2 years after the first dose of randomized study drug
  To compare the efficacy of two dose levels of L-Annamycin for Injection (190 versus 230 mg/m2/day) in combination with Cytarabine Injection (2.0 g/m2/day) versus placebo in combination with Cytarabine Injection as second line therapy for remission induction in adult subjects with refractory/relapsed AML as measured by overall survival (OS)
Part B - Confirmation of Efficacy of the Optimal Dosage Regimen as Measured by Overall Survival (OS) | From date of randomization to treatment (Day 1) to the date of death from any cause, assessed up to 2 years after the first dose of randomized study drug
  To confirm the efficacy of the optimal dosage regimen of L-Annamycin for Injection in combination with Cytarabine Injection (determined in Part A) versus placebo in combination with Cytarabine Injection as second line therapy for remission induction in adult subjects with refractory/relapsed AML as measured by OS;

CONTACTS AND LOCATIONS:
Locations (17):
- United States (2):
  - Bioresearch Partners, Miami, Florida
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
- Georgia (2):
  - GEORGIA: LLC ARENSIA Exploratory Medicine, Tbilisi
  - Caucasus Medical Center, Tbilisi
- RCCS Azienda Ospedaliero-Universitaria di Bologna, Istituto di Ematologia, Bologna, Italy
- LSMU Kauno klinikos, Kaunas, Lithuania
- Poland (5):
  - Szpital Kliniczny MSWiA z Warminsko-Mazurskim Centrum Onkologii w Olsztynie Oddział Kliniczny Hematologii i Chorób Wewnętrznych z Ośrodkiem Transplantacji Szpiku, Olsztyn
  - Oddział Hematologii i Transplantacji Szpiku, Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan
  - Uniwersytecki Szpital Kliniczny Klinika Hematologii i Transplantologii (Szczecin), Szczecin
  - Wojewódzki Szpital Zespolony im. L. Rydygiera w Toruniu, Oddział Hematologii, Torun
  - Instytut Hematologii i Transfuzjologii, Klinika Hematologii, Warsaw
- ARENSIA research clinic at the Oncology Institute "Prof. Dr. Ion Chiricuţă", Cluj-Napoca, Romania
- Spain (4):
  - Hospital Universitario Central de Asturias (HUCA), Oviedo, Principality of Asturias
  - Hospital MD Anderson Cancer Center Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario La Fe de Valencia, Valencia
- ARENSIA Exploratory Medicine, LLC, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided